CLINICAL TRIAL: NCT01412450
Title: DURABILITY-POP Study - Physician Initiated Trial Investigating the Efficacy of the Implant of Protégé EverFlex Nitinol Stents in Popliteal Lesions
Brief Title: Efficacity Study With the Protégé EverFlex Stent in Popliteal Lesions
Acronym: DUR-POP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Flanders Medical Research Program (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMRP-100702
Record Dates: First submitted 2010-07-02; First posted 2011-08-09 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Peripheral Arterial Disease
Keywords: symptomatic popliteal artery stenosis or occlusion
MeSH Terms: conditions — Peripheral Arterial Disease; Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nitinol stent (Experimental): Protégé EverFlex stent
  Interventions: Device: nitinol stent

INTERVENTIONS:
Device: nitinol stent — implantation of one Protégé EverFlex stent
  Other Names: Protégé EverFlex stent

SUMMARY:
This study will assess the results up to 12 months with the Protégé EverFlex stent (ev3) in patients presenting with a narrowing or blocking at the level of the knee artery, which leads to a limited walking distance, rest pain or non-healing ulcers.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion criteria

* De novo, restenotic or reoccluded lesion located in the popliteal artery, with or without superficial femoral artery involvement
* Patient presenting a score from 2 to 5 following Rutherford classification
* Patient is willing to comply with specified follow-up evaluations at the specified times
* Patient is >18 years old
* Patient (or their legal representative) understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
* Prior to enrollment, the guidewire has crossed target lesion
* Patient is eligible for treatment with the self-expanding nitinol EverFlex (ev3) stent

Angiographic Inclusion Criteria

* The target lesion has angiographic evidence of stenosis or restenosis > 50% or occlusion which can be passed with standard guidewire manipulation
* The target lesion, visually estimated, has a maximal length of 14 cm and can be categorized as either a type A or B lesions according the TASC II guidelines
* Target vessel diameter visually estimated is >3.5mm and <7.5 mm
* There is angiographic evidence of at least one-vessel-runoff to the foot

Exclusion Criteria:

* Presence of another stent in the target vessel that was placed during a previous procedure
* Presence of an aortic thrombosis or significant common femoral ipsilateral stenosis
* Previous by-pass surgery in the same limb
* Patients for whom antiplatelet therapy, anticoagulants or thrombolytic drugs are contraindicated
* Patients who exhibit persistent acute intraluminal thrombus of the proposed lesion site
* Perforation at the angioplasty site evidenced by extravasation of contrast medium
* Patients with known hypersensitivity to nickel-titanium
* Patients with uncorrected bleeding disorders
* Aneurysm located at the level of the SFA and/or popliteal artery
* Female patient with child bearing potential not taking adequate contraceptives or currently breastfeeding
* Life expectancy of less than twelve months
* Ipsilateral iliac treatment before the target lesion procedure with a residual stenosis > 30% or ipsilateral iliac treatment conducted after the target lesion procedure
* Use of thrombectomy, artherectomy or laser devices during procedure
* Any patient considered to be hemodynamically unstable at onset of procedure
* Patient is currently participating in another investigational drug or device study that has not completed the entire follow up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
primary patency | 12 months post-procedure
  primary patency at 12 months, defined as a target lesion without a hemodynamically significant stenosis on duplex ultrasound (systolic velocity ratio no greater than 2.4) and without TLR within 12 months

SECONDARY OUTCOMES:
Technical success | 1 day post-procedure
  Technical success, defined as the ability to cross and dilate the lesion to achieve residual angiographic stenosis no greater than 30% and residual stenosis less than 50% by duplex imaging
Primary patency rate at 6-, 12-month follow-up. | 6-, 12-month follow-up
  Patients that present without a hemodynamically significant stenosis at the target area on duplex ultrasound (systolic velocity ratio no greater than 2.4) and without prior TLR are defined as being primary patent.
Clinical success | 6-, 12-month follow-up
  Clinical success at follow-up is defined as an improvement of Rutherford classification at 6-, 12-month follow-up of one class or more as compared to the pre-procedure Rutherford classification.
tent fracture rate at 12-month follow-up | 12-month follow-up
  Determined according the following classification on x-ray: Class 0 (no strut factures); Class I (single tine fracture); Class II (multiple tine factures); Class III (Stent fracture(s) with preserved alignment of the components); Class IV (Stent fracture(s) with mal-alignment of the components); Class V (Stent fracture(s) in a trans-axial spiral configuration)
Serious adverse events | 1 year
  Defined as any clinical event that is fatal, life-threatening, or judged to be severe by the investigator; resulted in persistent or significant disability; necessitated surgical or percutaneous intervention; or required prolonged hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bosiers, MD, Principal Investigator — A.Z. Sint-Blasius
Locations (4):
- Belgium (4):
  - Imeldaziekenhuis, Bonheiden, Antwerp
  - University Hospital Antwerp, Edegem, Antwerp
  - A.Z. Sint-Blasius, Dendermonde, East-Flanders
  - Heilig-Hart Ziekenhuis, Tienen, Flemish Brabant